CLINICAL TRIAL: NCT04978311
Title: The Effects of Mirror Feedback Augmented Task-Specific and Impairment-Oriented Therapy With Home Practice in Stroke Rehabilitation
Brief Title: Mirror Feedback, Augmented Task-Specific, Impairment-Oriented Therapy, Home Practice, Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201812032RINA
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2022-08

CONDITIONS: Stroke Rehabilitation
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy (MT) priming with task-specific training (Experimental): In the regimen, participants will perform MT first followed by task-specific training. After completion of MT, participants will practice task-specific training that emphasizes on restoration of essential skills for daily activities. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Interventions: Behavioral: Mirror therapy (MT) priming with task-specific training
- Mirror therapy priming with impairment-oriented training (Active Comparator): In the regimen, participants will perform MT first followed by impairment-oriented training. After completion of MT, participants will practice impairment-oriented training that emphasizes on restoration of movement. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Interventions: Behavioral: Mirror therapy priming with impairment-oriented training
- Control therapy (Active Comparator): The control group will receive therapeutic training equivalent in duration to the two experimental groups. The control intervention will include practice of gross/fine motor activities, training of activities of daily living, practice to increase range of motions, muscle strengthening, as well as use of adaptive or compensatory technique to alleviate functional deficits. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Interventions: Behavioral: Control therapy

INTERVENTIONS:
Behavioral: Mirror therapy (MT) priming with task-specific training — In the regimen, participants will perform MT first followed by task-specific training. After completion of MT, participants will practice task-specific training that emphasizes on restoration of essential skills for daily activities. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Arms: Mirror therapy (MT) priming with task-specific training
Behavioral: Mirror therapy priming with impairment-oriented training — In the regimen, participants will perform MT first followed by impairment-oriented training. After completion of MT, participants will practice impairment-oriented training that emphasizes on restoration of movement. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Arms: Mirror therapy priming with impairment-oriented training
Behavioral: Control therapy — The control group will receive therapeutic training equivalent in duration to the two experimental groups. The control intervention will include practice of gross/fine motor activities, training of activities of daily living, practice to increase range of motions, muscle strengthening, as well as use of adaptive or compensatory technique to alleviate functional deficits. After that, the contents of home practice will be designed corresponding to treatment principles of the clinic-based intervention.
  Arms: Control therapy

SUMMARY:
In this study, the investigators will (1) examine immediate and long-term effects of MT priming with task-specific training versus MT-priming with impairment-oriented training, relative to a dose-matched control therapy on motor function, arm activities, quality of life, etc; (2) provide comprehensive evaluations based on the ICF model to identify the specific benefits of MT-priming regimens; and (3) explore demographic and clinical characteristics of participants that may predict treatment outcomes.

DETAILED DESCRIPTION:
Stroke is one of the major causes of long-term disability. Most stroke survivors suffer from arm paresis even in the chronic phase. There is a need to develop novel strategies to augment therapeutic efficacy in stroke rehabilitation. One potential method to enhance treatment efficacy is through the "priming" technique. Among all priming techniques, mirror therapy (MT) has been proposed to be a promising method to augment effects of motor re-training. The investigators propose a 3-year research project to determine the effects of MT-priming on augmenting stroke interventions. The investigators select two types of evidence-based neurorehabilitation, the task-specific training and the impairment-oriented training, to be primed by MT based on their unique treatment benefits on restoring arm ability. In addition, the investigators will provide customized home practice corresponding to each type of interventions. Specifically, the investigators will (1) examine immediate and long-term effects of MT priming with task-specific training versus MT-priming with impairment-oriented training, relative to a dose-matched control therapy on motor function, arm activities, quality of life, etc; (2) provide comprehensive evaluations based on the ICF model to identify the specific benefits of MT-priming regimens; and (3) explore demographic and clinical characteristics of participants that may predict treatment outcomes.

ELIGIBILITY:
Inclusion criteria:

* A first ever-stroke≧3 months
* Baseline Fugl-Meyer assessment of upper extremity scale (FMA-UE) between 18 to 56 (Fugl-Meyer et al. 1975)
* No excessive muscle spasticity of the affected arm (Modified Ashworth Scale < 3 at any joints of the affected arm) (Bohannon & Smith 1987)
* Able to follow examiners' commands and study instructions (Mini-Mental State Examination score≧22) (Folstein et al. 1975)
* No participation in any other experimental rehabilitation or drug studies during period of this project

Exclusion criteria:

* Concomitant neurologic, neuromuscular or orthopedic conditions that may interfere with participation of this project
* Epilepsy within three months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer Assessment (FMA) at 6 weeks, and 18 weeks | Baseline, 6 weeks, and 18 weeks
  The upper-extremity subscale of the FMA will be used to assess motor impairment. FMA contains 33 items (scale 0-66). The higher summed score means the greater recovery of motor impairment.
Change from Baseline Motor Activity Log (MAL) at 6 weeks, and 18 weeks | Baseline, 6 weeks and 18 weeks
  The MAL is a subjective outcome measure of an individual's real life functional upper limb performance. The MAL is administered by semi-structured interview to determine (a) how much (Amount of Use - AOU), and (b) how well the individual uses his upper limb (Quality of Movement - QOM) in real life.

SECONDARY OUTCOMES:
Change from Baseline Nottingham Extended Activities of Daily Living Scale (NEADL) at 6 weeks, and 18 weeks | Baseline, 6 weeks and 18 weeks
  The NEADL is a postal questionnaire to monitor the level of ADL disability in patients discharged into the community after rehabilitation. The tool assesses 21 activities within four categories: mobility, kitchen activities, domestic activities, and leisure activities. It provides an extended ADL score that is highly correlated with more complex, self-reported interviewer-administered measures of disability.
Change from Baseline Stroke Impact Scale Version 3.0 (SIS 3.0) at 6 weeks, and 18 weeks | Baseline, 6 weeks, and 18 weeks
  The SIS 3.0 is a stroke-specific health-related quality of life instrument. It consists of 59 items assessing 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation). Items are rated on a 5-point Likert scale, with lower scores indicating greater difficulty in task completion during the past week.
Change from Baseline Wolf Motor Function Test (WMFT) score at 6 weeks | Baseline and 6 weeks
  The WMFT quantifies the motor functions of the upper limbs through timed and functional tasks.
Change from Baseline Grip and Pinch strength at 6 weeks | Baseline and 6 weeks
  The Jamar Plus Digital Hand Dynamometer (Patterson Medical, Warrenville, IL, USA) was provided for measuring grip and pinch strength. Unilateral grip/pinch and bilateral grip/pinch are included.
Change from Baseline Chedoke Arm and Hand Activity Inventory (CAHAI) at 6 weeks | Baseline and 6 weeks
  The CAHAI measures arm and hand functions on 13 actual bilateral tasks on a 7-point scale (1 to 7). The properties of the CAHAI were studied, showing great interrater reliability and convergent and discriminant cross-sectional validity.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — School of Occupational Therapy, National Taiwan University, Taipei, Taiwan
Locations (2):
- Taiwan (2):
  - Feng Yuan Hospital, Taichung
  - National Taiwan University Hosipital, Taipei